CLINICAL TRIAL: NCT02101489
Title: Precise Transvaginal Tape Placement Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, M.D., Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206041
Record Dates: First submitted 2014-03-19; First posted 2014-04-02 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence
Keywords: TVT; Stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraop Foley catheter measurement (Active Comparator): 20 women will have intraoperative Foley catheter measurement of the urethral length
  Interventions: Other: Foley Catheter
- Without intraop Foley cath measurement (No Intervention): 20 women without intraoperative Foley catheter measurement of the urethral length

INTERVENTIONS:
Other: Foley Catheter — 20 with intraoperative Foley catheter measurement of the urethral length and 20 without
  Arms: Intraop Foley catheter measurement

SUMMARY:
This purpose of this study is to study is to see if intra-operative urethral length measurement with the Foley catheter will improve the placement of a synthetic sling in the mid-urethra.

DETAILED DESCRIPTION:
This study will assess the effect of intraoperative measurement of the urethral length with the Foley catheter in optimization of sling placement in the mid female urethra. Of note, the Foley catheter is well-tolerated, placed routinely during surgery to drain the bladder and has no complications associated with it. Women who have chosen to undergo trans-vaginal tape sling (TVT) for stress urinary incontinence will be asked to enroll in this randomized trial by the study team during their clinic visit. Randomization will be performed by the FPMRS study nurse coordinator after a woman has given her informed consent and meets the study criteria. Twenty women will be randomized to undergo measurement of the urethral length by marking the Foley catheter at the urethral meatus when it is placed at the start of the surgical case. When the catheter is removed, the length from the end of the Foley balloon to the marking at the urethra will be measured as urethral length, the mid urethral point will then be determined by dividing the urethral length be two where the incision of sling placement will be made and twenty women will have our usual pre-operative assessment (which does not include intraoperative measurement of the urethral length with the Foley catheter) for the treatment of symptomatic stress urinary incontinence All women participating in the study will receive an intra-operative 3-D trans-vaginal ultrasound (BK Flex Focus ultrasound with the 8838 transvaginal probe). The image will be stored and reviewed for; urethral length, urethral sphincter complex length and width. All women in the study will have an ultrasound at the end of their surgical procedure and a follow-up ultrasound at 2 weeks post operatively to assess for sling migration. Of note, transvaginal ultrasound is well-tolerated and has no complications associated with it. All ultrasound measurements will be done by a four qualified surgeons, Dr. Elizabeth Mueller Dr. Ahmed Akl, Dr. Tanaka Dune, and Dr. Susanne Taege who have been trained on ultrasound measurements. In addition, women will complete questionnaires assessing their pelvic floor symptoms pre-operatively and at 2 week following surgery. Instruments used will be the Pelvic Floor Disorders Inventory (PFDI), Medical Epidemiologic and Social Aging (MESA) and the Patient Global Impression of Improvement (PGII) [11, 12].

ELIGIBILITY:
Inclusion Criteria:

* Candidates for TVT
* >=18 years of age to participate

Exclusion Criteria:

* Inability to give informed consent
* Previous SUI(stress urinary incontinence) treatment including TVT, Burch or urethral bulking agents
* Previous bladder, urethral malignancies or vaginal/pelvic radiation treatment.
* Pregnant women cannot participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
If using a Foley catheter is a reliable way to measure the urethral length before placing the tension free vaginal tape in the mid-urethra. | 2 weeks
  measurement of the urethral length by marking the Foley catheter at the urethral meatus when it is placed at the start of the surgical case. When the catheter is removed, the length from the end of the Foley balloon to the marking at the urethra will be measured as urethral length, the mid urethral point will then be determined by dividing the urethral length be two where the incision of sling placement will be made.

SECONDARY OUTCOMES:
Comparing urethral length measurement with the Foley catheter and 3D ultrasound. | 2 weeks
  All women in the study will have an ultrasound at the end of their surgical procedure and a follow-up ultrasound at 2 weeks post operatively to assess for sling migration.
Location change of mid-urethral slings from the time of surgery to 2 weeks after surgery. | 2 weeks
  We will then compare the mid-point location of the midurethral sling between the group that received an intra-op Foley catheter measurement to the group that didn't receive the Foley catheter.
Stratify the data based on patient race, BMI, prolapse and age | 6 weeks
  Stratify the data based on patient race, BMI, prolapse and age

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Mueller, M.D., Principal Investigator — Loyola University
Locations (1):
- Loyola University Health System, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aigmueller T, Trutnovsky G, Tamussino K, Kargl J, Wittmann A, Surtov M, Kern P, Frudinger A, Riss P, Bjelic-Radisic V. Ten-year follow-up after the tension-free vaginal tape procedure. Am J Obstet Gynecol. 2011 Nov;205(5):496.e1-5. doi: 10.1016/j.ajog.2011.07.010. Epub 2011 Jul 20. PMID 21944223
- [Background] Olsson I, Abrahamsson AK, Kroon UB. Long-term efficacy of the tension-free vaginal tape procedure for the treatment of urinary incontinence: a retrospective follow-up 11.5 years post-operatively. Int Urogynecol J. 2010 Jun;21(6):679-83. doi: 10.1007/s00192-009-1083-7. Epub 2010 Jan 13. PMID 20069417
- [Background] Nilsson CG, Palva K, Rezapour M, Falconer C. Eleven years prospective follow-up of the tension-free vaginal tape procedure for treatment of stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1043-7. doi: 10.1007/s00192-008-0666-z. Epub 2008 Jun 6. PMID 18535753
- [Background] Nilsson CG, Palva K, Aarnio R, Morcos E, Falconer C. Seventeen years' follow-up of the tension-free vaginal tape procedure for female stress urinary incontinence. Int Urogynecol J. 2013 Aug;24(8):1265-9. doi: 10.1007/s00192-013-2090-2. Epub 2013 Apr 6. PMID 23563892
- [Background] Bjelic-Radisic V, Dorfer M, Greimel E, Frudinger A, Tamussino K, Winter R. Quality of life and continence 1 year after the tension-free vaginal tape operation. Am J Obstet Gynecol. 2006 Dec;195(6):1784-8. doi: 10.1016/j.ajog.2006.07.014. PMID 17132481
- [Background] Kociszewski J, Rautenberg O, Perucchini D, Eberhard J, Geissbuhler V, Hilgers R, Viereck V. Tape functionality: sonographic tape characteristics and outcome after TVT incontinence surgery. Neurourol Urodyn. 2008;27(6):485-90. doi: 10.1002/nau.20556. PMID 18288705
- [Background] Rahn DD, Marinis SI, Schaffer JI, Corton MM. Anatomical path of the tension-free vaginal tape: reassessing current teachings. Am J Obstet Gynecol. 2006 Dec;195(6):1809-13. doi: 10.1016/j.ajog.2006.07.009. PMID 17132484
- [Background] McGuire EJ, Lytton B. Pubovaginal sling procedure for stress incontinence. 1978. J Urol. 2002 Feb;167(2 Pt 2):1120-3; discussion 1124. doi: 10.1016/s0022-5347(02)80355-x. No abstract available. PMID 11905885
- [Background] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495